CLINICAL TRIAL: NCT06344442
Title: Effect of Low-dose Arginine-vasopressin Supplementation on Post-transplant Acute Kidney Injury After Liver Transplantation
Brief Title: Low-dose Arginine-vasopressin Supplementation on Post-transplant Acute Kidney Injury After Liver Transplantation (AVENIR Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220827
Record Dates: First submitted 2024-02-23; First posted 2024-04-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury Post Liver Transplantation
Keywords: Low dose arginine -vasopressin Acute Kidney injury Liver transplantation
MeSH Terms: interventions — Arginine Vasopressin; Norepinephrine

STUDY DESIGN:
Intervention Model Description: Prospective, national multicentre, double-blinded, randomized ,controlled superiority trial with two parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the clinical teams involved intraoperatively (anaesthetists, nurse anaesthetists and surgeons) and postoperatively (doctors and nurses who will take care of the patient postoperatively) and the families will ignore the allocation of treatments for the duration of the trial,except the nurse in charge of preparing the infusions ,She will ensure respect for the blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arginine vasopressin (Experimental): low-dose arginine-vasopressin supplementation group: Vasopressin will be administered by continuous infusion. AVP will be used to a final concentration of 0.12 U/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that AVP doses ranged from 0.01 to 0.06 U/min
  Interventions: Drug: Arginine vasopressin
- Norepinephrine (Active Comparator): Norepinephrine will be administered by continuous infusion. Norepinephrine will be used with final concentrations of 120 microg/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that NE doses ranged from10 to 60 microg/min.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Arginine vasopressin — low-dose arginine-vasopressin supplementation group: Vasopressin will be administered by continuous infusion. AVP will be used to a final concentration of 0.12 U/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that AVP doses ranged from 0.01 to 0.06 U/min.
  Arms: Arginine vasopressin
Drug: Norepinephrine — Norepinephrine will be administered by continuous infusion. Norepinephrine will be used with final concentrations of 120 microg/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that NE doses ranged from10 to 60 microg/min.
  Arms: Norepinephrine

SUMMARY:
Liver transplantation (LT) is a high-risk surgery for hemodynamic instability and haemorrhagic shock with a high-risk of acute kidney injury (AKI). Indeed, the incidence of post-transplant AKI exceeds 50% in some series with 15% of patients requiring renal replacement therapy. Acute kidney injury after LT is a predisposing factor for chronic renal failure which is independently associated with higher morbidity and mortality.

Arginine vasopressin (AVP), an essential stress hormone released in response to hypotension, binds to AVPR1a to promote vasoconstriction. Furthermore, it may have nephroprotective effects with a preferential vasoconstriction of the post-glomerular arteriole resulting in increased glomerular filtration

The hypothesis of the present work is that low-dose arginine-vasopressin supplementation reduce posttransplant AKI in liver transplantation.

DETAILED DESCRIPTION:
Prospective, national multicenter, double-blinded, randomized , controlled superiority trial with two parallel arms : AVP vs Norepinephrine

The primary objective is to demonstrate that intraoperative low-dose supplementation of AVP induces a reduction in posttransplant AKI after liver transplantation

Investigational medicinal product: vasopressin will be administered by continuous infusion. AVP will be used to a final concentration of 0.12 U/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that AVP doses ranged from 0.01 to 0.06 U/min.

Comparator treatment : norepinephrine will be administered by continuous infusion. Norepinephrine will be used with final concentrations of 120 microg/ml. The vasopressor infusion will be titrated to maintain an MAP of at least 65 mmHg. The study-drug infusion will be started at 5 ml/h and increased by 2.5 ml/h to achieve a maximum target rate of 30 ml/h, so that NE doses ranged from10 to 60 microg/min.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any adult patient with a scheduled liver transplantation
* All participants will need to be given clear information about the study and give signed informed consent.
* Person affiliated to the Social Security

Exclusion Criteria:

* Super-emergency for liver transplantation or fulminant hepatitis
* Patient listed for or receiving simultaneous liver-kidney transplantation (SLKT)
* Patients with end-stage renal disease (chronic eGFR < 15 mL/min/1.73 m2 or requiring extra-renal purification before liver transplantation
* Patient with epilepsy
* Hypersensitivity to arginine-vasopressin and to its excipients
* Patient refusal
* Patients for whom it is impossible to give informed consent (language barrier)
* Adults under guardianship or trusteeship, persons deprived of their liberty
* Patient enrolled in another interventional clinical study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare the effect of intraoperative low-dose supplementation of AVP vs norepinephrine infusions on post-transplant Acute Kidney Injury after liver transplantation. | during the first 7 postoperative days
  The stages of AKI according to AKI Network criteria (KDIGO score) determined by changes in serum creatinine and changes in urine output.

SECONDARY OUTCOMES:
To compare into the two arms the number of packed red blood cellsand fresh frozen plasma transfused | during the first 12 hours postoperatively
To compare into the two arms the number of the Number of AKI KDIGO 1 | 1 during the first 7days
  defined as increase in serum creatinine concentration by 1.5 to 1.9 fold or ≥0.3mg/dl (or 27 micromol/L) within 48h or urine output <0.5 ml/Kg/h over a period 6-12 h)
To compare into the two arms the Number of AKI KDIGO 2 | during the first 7 postoperative
  defined as increase in serum creatinine concentration by 2.0 to 2.9 fold or urine output <0.5 ml/Kg/h over a period ≥12 h)
To compare into the Number of AKI KDIGO 3 | during the first 7 postoperative
  defined as increase in serum creatinine concentration ≥ 3 fold or ≥ 4mg/dl (or 354 micromol/L) or urine output <0.3 ml/Kg/h for ≥24h or anuria>12h)
The need for renal replacement for replacement therapy (RRT) in ICU | during the first 7 days postoperatively and on postoperative day 30
The number of patients remaining on dialysis at the end of the study | on the 30th Day
Average intraoperative norepinephrine concentrations | intraoperative
Average intraoperative concentrations of other vasopressors and inotropes (Adrenalin, Dobutamine) | intraoperative
Number of platelets transfused intraoperatively | during the first 12 hours postoperatively.
Amount of vascular filling solutions intraoperatively | During the first 12 hours postoperatively.
Sequential Organ Failure Assessment (SOFA score) | On the third and seventh postoperative day
  Sequential Organ Failure Assessment (SOFA score between 0 and 24). Zero indicates that the patient has no organ dysfunction, twenty-four is the maximum score and indicates that the patient has vinght four is the maximum score and indicates that the patient has all 6 of the organ dysfunctions explored.
  (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic)
Number of days alive outside intensive care unit | during the 30 day post-operation
Mortality | at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DURANTEAU, Pr, Study Director — Département Anesthésie-Réanimation - Université Paris-Saclay Hospital Bicêtre - Paul Brousse; Gilles LEBUFFE, Pr, Principal Investigator — Service Anesthésie-Réanimation - CHU de Lille; Daniel EYRAUD, Pr, Principal Investigator — Service Anesthésie-Réanimation -APHP Pitié-Salpêtrière; Emmanuel WEISS, Pr, Principal Investigator — Service Anesthésie-Réanimation - APHP hôpital Beaujon; Antoine DEWITTE, Pr, Principal Investigator — Service Anesthésie-Réanimation -CHU de Bordeaux centre médicochirurgical Magellan hôpital Haut Lévêque; Baptiste LORDIER, Pr, Principal Investigator — Service Anesthésie-Réanimation -CHU de Strasbourg Hôpital de Hautepierre; Alice BLET, Pr, Principal Investigator — Service Anesthésie-Réanimation - Hôpital de la Croix Rousse
Locations (1):
- URC Lariboisière-Fernand Widal-saint Louis, Paris, France

REFERENCES:
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Hilmi IA, Damian D, Al-Khafaji A, Planinsic R, Boucek C, Sakai T, Chang CC, Kellum JA. Acute kidney injury following orthotopic liver transplantation: incidence, risk factors, and effects on patient and graft outcomes. Br J Anaesth. 2015 Jun;114(6):919-26. doi: 10.1093/bja/aeu556. Epub 2015 Feb 10. PMID 25673576
- [Result] Watt KD, Pedersen RA, Kremers WK, Heimbach JK, Charlton MR. Evolution of causes and risk factors for mortality post-liver transplant: results of the NIDDK long-term follow-up study. Am J Transplant. 2010 Jun;10(6):1420-7. doi: 10.1111/j.1600-6143.2010.03126.x. Epub 2010 May 10. PMID 20486907
- [Result] Hajjar LA, Vincent JL, Barbosa Gomes Galas FR, Rhodes A, Landoni G, Osawa EA, Melo RR, Sundin MR, Grande SM, Gaiotto FA, Pomerantzeff PM, Dallan LO, Franco RA, Nakamura RE, Lisboa LA, de Almeida JP, Gerent AM, Souza DH, Gaiane MA, Fukushima JT, Park CL, Zambolim C, Rocha Ferreira GS, Strabelli TM, Fernandes FL, Camara L, Zeferino S, Santos VG, Piccioni MA, Jatene FB, Costa Auler JO Jr, Filho RK. Vasopressin versus Norepinephrine in Patients with Vasoplegic Shock after Cardiac Surgery: The VANCS Randomized Controlled Trial. Anesthesiology. 2017 Jan;126(1):85-93. doi: 10.1097/ALN.0000000000001434. PMID 27841822
- [Result] Pecci A, Balduini CL. Desmopressin and super platelets. Blood. 2014 Mar 20;123(12):1779-80. doi: 10.1182/blood-2014-01-551242. No abstract available. PMID 24652962
- [Result] Sims CA, Holena D, Kim P, Pascual J, Smith B, Martin N, Seamon M, Shiroff A, Raza S, Kaplan L, Grill E, Zimmerman N, Mason C, Abella B, Reilly P. Effect of Low-Dose Supplementation of Arginine Vasopressin on Need for Blood Product Transfusions in Patients With Trauma and Hemorrhagic Shock: A Randomized Clinical Trial. JAMA Surg. 2019 Nov 1;154(11):994-1003. doi: 10.1001/jamasurg.2019.2884. PMID 31461138
- [Result] Okazaki N, Iguchi N, Evans RG, Hood SG, Bellomo R, May CN, Lankadeva YR. Beneficial Effects of Vasopressin Compared With Norepinephrine on Renal Perfusion, Oxygenation, and Function in Experimental Septic Acute Kidney Injury. Crit Care Med. 2020 Oct;48(10):e951-e958. doi: 10.1097/CCM.0000000000004511. PMID 32931198
- [Result] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Result] Gordon AC, Russell JA, Walley KR, Singer J, Ayers D, Storms MM, Holmes CL, Hebert PC, Cooper DJ, Mehta S, Granton JT, Cook DJ, Presneill JJ. The effects of vasopressin on acute kidney injury in septic shock. Intensive Care Med. 2010 Jan;36(1):83-91. doi: 10.1007/s00134-009-1687-x. Epub 2009 Oct 20. PMID 19841897
- [Result] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Result] Edwards RM, Trizna W, Kinter LB. Renal microvascular effects of vasopressin and vasopressin antagonists. Am J Physiol. 1989 Feb;256(2 Pt 2):F274-8. doi: 10.1152/ajprenal.1989.256.2.F274. PMID 2916660
- [Result] Holmes CL, Patel BM, Russell JA, Walley KR. Physiology of vasopressin relevant to management of septic shock. Chest. 2001 Sep;120(3):989-1002. doi: 10.1378/chest.120.3.989. PMID 11555538
- [Result] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211